CLINICAL TRIAL: NCT06042387
Title: Genome Analysis Across Populations in Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mark Silverberg, Dr., Mount Sinai Hospital, Canada
Other Study IDs: 02-0234-E; U01DK062423 (NIH)
Record Dates: First submitted 2023-05-31; First posted 2023-09-18 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis; Healthy; Crohn Disease; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participation involves:
  One-time blood (preferred) or saliva sample Collection of clinical data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IBD Subjects: Available medical records to confirm IBD diagnosis (Crohn's disease, Ulcerative colitis, IBD undetermined (IBD-U)) Any age Willing to provide blood or saliva sample
  Interventions: Genetic: Blood or saliva sample collection
- Controls: No personal history of IBD, no family history of IBD, no history of unexplained chronic diarrhea/blood in stool/anemia/abdominal pain/weight loss Any age Willing to provide blood or saliva sample
  Interventions: Genetic: Blood or saliva sample collection

INTERVENTIONS:
Genetic: Blood or saliva sample collection — Blood or saliva sample & clinical data collection

SUMMARY:
Objective:

To use clinical, genetic and genome analysis to better understand and define the genetic and environmental factors that contribute to IBD within affected populations.

DETAILED DESCRIPTION:
Background:

Inflammatory bowel disease (IBD) is a chronic, and often disabling, disorder of the intestines characterized by dysregulation of mucosal immune response. Recent data suggests that the incidence and prevalence rates among all populations may be increasing due to constantly changing environmental exposures. The goal of the study is to identify susceptible genes that contribute to the pathogenesis of IBD in affected individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects: diagnosed with Inflammatory Bowel Disease (Crohn's disease, ulcerative colitis, IBD-undetermined)
* Available medical records to confirm IBD diagnosis (Crohn's disease, Ulcerative colitis, IBD undetermined (IBD-U))
* Healthy controls: no personal history of IBD, no family history of IBD, no history of unexplained chronic diarrhea/blood in stool/anemia/abdominal pain/weight loss
* Any age

Exclusion Criteria:

- Subjects with other gastrointestinal conditions not meeting the above IBD or Healthy Control criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: IBD or Healthy controls (non-IBD)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Genomics studies across populations | 2022-2027
  Whole Exome Sequencing (+/- other sequencing) is planned

CONTACTS AND LOCATIONS:
Overall Officials: Mark Silverberg, MD PhD, Principal Investigator — Sinai Health System
Locations (1):
- Sinai Health System, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided